CLINICAL TRIAL: NCT00479284
Title: Contribution of Average Volume Assured Pressure Support (AVAPS) to Efficacy of bi-Level Pressure Support Nocturnal Ventilation and Impact on Sleep Structure
Brief Title: Efficacy of Average Volume Assured Pressure Support With Bi-Level Pressure Support Nocturnal Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ligue Pulmonaire Genevoise (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Protocol 06-094
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Hypercapnic Respiratory Failure; Obesity Hypoventilation Syndrome; Chronic Obstructive Pulmonary Disease
Keywords: Non-invasive ventilation; Polysomnography; Average volume assured pressure support
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Average volume assured pressure support (AVAPS)

SUMMARY:
Patients with chronic hypercapnic respiratory failure can be successfully treated with home nocturnal non-invasive ventilation. Bi-level pressure support ventilators are at present the most frequently used ventilators for long term home ventilation. A recently commercialized bi-level ventilator offers the feature of automatically adjusting pressure support on the basis of a pre-determined ideal effective ventilation. Because this option may induce important swings in pressure support, and thus patient discomfort, and maybe increase leaks, we chose to analyse the impact of average volume assured pressure support (AVAPS) on patient comfort, subjective and objective quality of sleep and efficacy of ventilatory support.

DETAILED DESCRIPTION:
This study aims to compare, in a randomized order, two consecutive nights with a bi-level positive pressure ventilator (Synchrony, Respironics, USA), with and without average volume assured pressure support (AVAPS), in patients with chronic respiratory failure, treated on a long term basis by home nocturnal non-invasive ventilation.

Specific endpoints are :

* quality of sleep assessed by polysomnography scored by an independent investigator (sleep efficiency, distribution of sleep stages, arousals and sleep stage changes) and subjective scores (St Mary's questionnaire),
* perception of comfort of ventilation (clinical score),
* efficacy of ventilation (pulsoximetry, transcutaneous capnography (Tina TCM4 Radiometer, Copenhagen), effective ventilation and tidal volumes, leaks as measured by ventilator, Stardust software, Respironics).

Patients: Fourteen patients with obesity-hypoventilation and/or COPD, treated and stable for at least 3 months, will be included and undergo complete sleep studies in Geneva University Hospital's Sleep Laboratory. Patients included must be compliant to treatment (at least 4 hours of use of ventilator/night).

Methods: Patients are blinded as to whether or not AVAPS is implemented. Target tidal volume is set at 7-8 ml/kg. EPAP (Expiratory positive airway pressure) level is unchanged. Minimal IPAP (Inspiratory positive airway pressure) level is set at usual IPAP - 3 cm H2O. Maximal IPAP is set between 25 and 30 cm H2O. Back up frequency is unchanged.

All patients must provide written informed consent. Protocol has been accepted by the ethics committee on clinical research of Geneva University Hospital.

Results of scores, and relevant parameters of polysomnography, oxymetry, and capnography, will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for chronic hypercapnic respiratory failure by home bi-level positive pressure non-invasive ventilation for at least 3 months, in a stable clinical condition

Exclusion Criteria:

* Poor compliance (< 4 hours/day) to home ventilation or recent episode ( < 3 months) of cardiac or respiratory failure necessitating hospitalization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-06; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Quality of sleep | One night
Efficacy of ventilation | One night

SECONDARY OUTCOMES:
Patient comfort | One night

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, M.D., Principal Investigator — Division of Lung Diseases, Department of Medicine, Geneva University Hospital
Locations (1):
- Sleep Laboratory; Department of Psychiatry, Geneva University Hospital, Chêne-Bourg, Canton of Geneva, Switzerland